CLINICAL TRIAL: NCT02102360
Title: Conventional or Minimally Invasive Surgical Technique for the Treatment of Furcation Defects Using Enamel Matrix Derivative and Anorganic Bovine Bone - a Randomized Controlled Clinical Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tulio Bonna Pignaton, Conventional or minimally invasive surgical technique for the treatment of furcation defects using enamel matrix derivative and anorganic bovine bone - a randomized controlled clinical trial., University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Mist2014
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Furcation Defects; Periodontal Disease
Keywords: microsurgery, furcation defects, periodontal disease, enamel matrix proteins, bone substitutes
MeSH Terms: conditions — Furcation Defects; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Minimally invasive surgical technique (MIST) (Experimental): A minimally invasive surgical technique was performed to access mandibular furcation defects in the test group, aiming to perform minimal flap reflection, minimal wound, and gentle handling of the soft and hard tissue in periodontal surgery. The use of a microsurgical approach provides magnification and optimal illumination of the surgical site improving visual acuity. Further advantages may be the reduction of flap reflection during surgery, consequently advantages in wound healing process and benefits in patient's perceptions of the procedure. A less invasive surgical procedure may lead to a less cell demand in the healing process, and a potentially reduced morbidity. The minimally invasive surgical procedures were performed using microscope.
  Interventions: Device: Anorganic Bovine Bone; Device: Enamel Matrix Derivative
- Conventional surgical technique (CST) (Experimental): A conventional surgical technique was performed to access mandibular furcation defects in the control group.
  Interventions: Device: Anorganic Bovine Bone; Device: Enamel Matrix Derivative

INTERVENTIONS:
Device: Anorganic Bovine Bone — used to improve periodontal regenerative procedures.
  Other Names: Anorganic Bovine Bone (Bio-Oss, Geistlich Pharma).
Device: Enamel Matrix Derivative — used to improve periodontal regenerative procedures.
  Other Names: Enamel Matrix Derivative (Emdogain - Institute Straumann, Switzerland).

SUMMARY:
This clinical study compared a conventional surgical technique (CST) and a minimally invasive surgical technique (MIST) in the regenerative treatment of mandibular furcation defects.

DETAILED DESCRIPTION:
Using a split-mouth design, fifteen patients with bilateral class II and III furcation defects were treated with MIST (Test Group) or CST (Control Group). Furcation defects in both groups were filled with anorganic bovine bone (ABB) and enamel matrix derivative (EMD). Patient-centered outcomes including analyses of pain, discomfort, edema, hematoma, root hypersensitivity and daily activities interference were recorded using a Visual Analogue Scale seven days after surgeries. Clinical and radiographic parameters were assessed at baseline and 6 months postoperatively. Data were statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

(I) subjects with a diagnosis of periodontitis; (II) presence of one pair of contralateral mandibular molars with buccal / lingual furcation defects; (III) non-smokers; (IV) plaque index < 20%.

Exclusion Criteria:

(I) patients that presented systemic disease; (II) had taken antibiotics in the past 6 months prior to surgery; (III) pregnant women or lactating mothers; (IV) molars with periapical disease; (V) cervical restorations or prosthesis closer than 1 mm to fornix; (VI) lingual furcation defects presenting gingival recession (GR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Horizontal clinical attachment level (HCAL) | baseline and 6 months after surgical procedure
  The clinical measure HCAL was assessed and recorded by an experienced periodontist, blinded to the procedures to assess the efficacy of surgical procedures.

SECONDARY OUTCOMES:
Pain Scores on the Visual Analogue Scale | 7 days after surgery
Discomfort Scores on the Visual Analogue Scale | 7 days after surgery
Edema Scores on the Visual Analogue Scale | 7 days after surgery
Hematoma Scores on the Visual Analogue Scale | 7 days after surgery
Root Hypersensitivity Scores on the Visual Analogue Scale | 7 days after surgery
Daily Activities Interference Scores on the Visual Analogue Scale | 7 days after surgery
Vertical clinical attachment level (VCAL) | baseline and 6 months
  The clinical measure HCAL was assessed and recorded by an experienced periodontist, blinded to the procedures to assess the efficacy of surgical procedures.
Probing pocket depth (PPD) | baseline and 6 months
  The clinical measure HCAL was assessed and recorded by an experienced periodontist, blinded to the procedures to assess the efficacy of surgical procedures
Gingival recession | baseline and 6 months
  The clinical measure HCAL was assessed and recorded by an experienced periodontist, blinded to the procedures to assess the efficacy of surgical procedures

OTHER OUTCOMES:
Digital subtraction radiography density gain | baseline and 6 months
  The radiographs were obtained with the paralleling technique employing an x-ray unit and a digital sensor . Customized radiographic holders for each patient . Digital subtraction radiographs (DSR) were performed using a specific software. All pairs of baseline and 6-month radiographs for each treated site were then subtracted.
  Standardized regions of interest (ROIs) were select for each subtracted digital image: (1) placed in the bone's most coronal and central aspect of the furcation defect; and (2) placed at a distant untreated site acting as a radiographic control. The ROIs were not superimposed on any portion of the tooth surface. A software (Image Tool for Windows, Version 3.0, USA) was used to assess radiographic density changes that occurred in ROIs.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral & Maxillofacial Surgery and Periodontology, School of Dentistry of Ribeirao Preto, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Cortellini P, Tonetti MS. Microsurgical approach to periodontal regeneration. Initial evaluation in a case cohort. J Periodontol. 2001 Apr;72(4):559-69. doi: 10.1902/jop.2001.72.4.559. PMID 11338311
- [Background] Cortellini P, Tonetti MS. A minimally invasive surgical technique with an enamel matrix derivative in the regenerative treatment of intra-bony defects: a novel approach to limit morbidity. J Clin Periodontol. 2007 Jan;34(1):87-93. doi: 10.1111/j.1600-051X.2006.01020.x. PMID 17243998
- [Background] Cortellini P, Tonetti MS. Minimally invasive surgical technique and enamel matrix derivative in intra-bony defects. I: Clinical outcomes and morbidity. J Clin Periodontol. 2007 Dec;34(12):1082-8. doi: 10.1111/j.1600-051X.2007.01144.x. Epub 2007 Oct 22. PMID 17953696
- [Background] Cortellini P, Tonetti MS. Focus on intrabony defects: guided tissue regeneration. Periodontol 2000. 2000 Feb;22:104-32. doi: 10.1034/j.1600-0757.2000.2220108.x. No abstract available. PMID 11276509
- [Background] Cortellini P, Prato GP, Tonetti MS. The modified papilla preservation technique. A new surgical approach for interproximal regenerative procedures. J Periodontol. 1995 Apr;66(4):261-6. doi: 10.1902/jop.1995.66.4.261. PMID 7782979
- [Background] Wang HL, Greenwell H, Fiorellini J, Giannobile W, Offenbacher S, Salkin L, Townsend C, Sheridan P, Genco RJ; Research, Science and Therapy Committee. Periodontal regeneration. J Periodontol. 2005 Sep;76(9):1601-22. doi: 10.1902/jop.2005.76.9.1601. PMID 16171453
- [Background] Tsao YP, Neiva R, Al-Shammari K, Oh TJ, Wang HL. Factors influencing treatment outcomes in mandibular Class II furcation defects. J Periodontol. 2006 Apr;77(4):641-6. doi: 10.1902/jop.2006.050133. PMID 16584345
- [Background] Martin M, Gantes B, Garrett S, Egelberg J. Treatment of periodontal furcation defects. (I). Review of the literature and description of a regenerative surgical technique. J Clin Periodontol. 1988 Apr;15(4):227-31. doi: 10.1111/j.1600-051x.1988.tb01575.x. PMID 3290276
- [Background] Hammarstrom L, Heijl L, Gestrelius S. Periodontal regeneration in a buccal dehiscence model in monkeys after application of enamel matrix proteins. J Clin Periodontol. 1997 Sep;24(9 Pt 2):669-77. doi: 10.1111/j.1600-051x.1997.tb00248.x. PMID 9310871
- [Background] Hammarstrom L. Enamel matrix, cementum development and regeneration. J Clin Periodontol. 1997 Sep;24(9 Pt 2):658-68. doi: 10.1111/j.1600-051x.1997.tb00247.x. PMID 9310870
- [Background] Heijl L. Periodontal regeneration with enamel matrix derivative in one human experimental defect. A case report. J Clin Periodontol. 1997 Sep;24(9 Pt 2):693-6. doi: 10.1034/j.1600-051x.1997.00693.x. PMID 9310874
- [Background] Dori F, Arweiler NB, Szanto E, Agics A, Gera I, Sculean A. Ten-year results following treatment of intrabony defects with an enamel matrix protein derivative combined with either a natural bone mineral or a beta-tricalcium phosphate. J Periodontol. 2013 Jun;84(6):749-57. doi: 10.1902/jop.2012.120238. Epub 2012 Aug 8. PMID 22873657
- [Background] Tonetti MS, Fourmousis I, Suvan J, Cortellini P, Bragger U, Lang NP; European Research Group on Periodontology (ERGOPERIO). Healing, post-operative morbidity and patient perception of outcomes following regenerative therapy of deep intrabony defects. J Clin Periodontol. 2004 Dec;31(12):1092-8. doi: 10.1111/j.1600-051X.2004.00615.x. PMID 15560811
- [Background] Polimeni G, Xiropaidis AV, Wikesjo UM. Biology and principles of periodontal wound healing/regeneration. Periodontol 2000. 2006;41:30-47. doi: 10.1111/j.1600-0757.2006.00157.x. No abstract available. PMID 16686925